CLINICAL TRIAL: NCT03214120
Title: Does Modified Ultrafiltration Affect Thromboelastography Results?
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: K5900405
Record Dates: First submitted 2017-07-04; First posted 2017-07-11 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Congenital Heart Disease
Keywords: thromboelastography, modified ultrafiltration
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is to evaluate the effect of modified ultrafiltration on different components of Thromboelastography (TEG) in neonates undergoing cardiac surgery using cardiopulmonary bypass.

DETAILED DESCRIPTION:
The study will be performed at Advocate Children's Hospital, Oak Lawn. All neonates undergoing cardiac operations with cardiopulmonary bypass and modified ultrafiltration will be enrolled. Parents will be consented before surgery.

After weaning from cardiopulmonary bypass and before starting modified ultrafiltration, a TEG sample will be taken. The components studied are Reaction time (R), Coagulation time (K), Angle, Maximum Amplitude (MA) and whole blood clot lysis index at 30 minutes (LY30). Another TEG sample will be taken after finishing modified ultrafiltration and before protamine is given. The different components will be compared pre and after modified ultrafiltration. The Primary end points are the changes of the different TEG components after modified ultrafiltration. The secondary end points are the utilization of different blood products (packed red cells, fresh frozen plasma and platelets transfusion) during and after surgery.

ELIGIBILITY:
Inclusion Criteria: - neonates

* congenital heart disease
* pediatric cardiac operation with cardiopulmonary bypass
* modified ultrafiltration done at the end of cardiopulmonary bypass

Exclusion Criteria: -patients older than 1 month.

* Cardiopulmonary bypass is not used
* Modified ultrafiltration is not performed

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates with congenital heart disease requiring cardiac surgery during the first month of life, with the use of cardiopulmonary bypass and modified ultrafiltration.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
change in thromboelastography components after modified ultrafiltration | 1 hour (time during surgery after doing modified ultrafiltration) to 2 days (postoperative recovery in intensive care unit)
  effect of modified ultrafiltration on different components of thromboelastography

SECONDARY OUTCOMES:
blood products utilization during and after surgery | initial phase of recovery (2 days) in the intensive care unit after cardiac surgery
  use of packed red cells, fresh frozen plasma and platelets during or after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chawki Elzein, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Advocate Children's Hospital, Oak Lawn, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moat NE, Rebuck N, Shore DF, Evans TW, Finn AH. Humoral and cellular activation in a simulated extracorporeal circuit. Ann Thorac Surg. 1993 Dec;56(6):1509-14. doi: 10.1016/0003-4975(93)90742-z. PMID 7505562
- [Result] Luciani GB, Menon T, Vecchi B, Auriemma S, Mazzucco A. Modified ultrafiltration reduces morbidity after adult cardiac operations: a prospective, randomized clinical trial. Circulation. 2001 Sep 18;104(12 Suppl 1):I253-9. doi: 10.1161/hc37t1.094931. PMID 11568065
- [Result] Kane LC, Woodward CS, Husain SA, Frei-Jones MJ. Thromboelastography--does it impact blood component transfusion in pediatric heart surgery? J Surg Res. 2016 Jan;200(1):21-7. doi: 10.1016/j.jss.2015.07.011. Epub 2015 Jul 10. PMID 26237992
- [Result] Niebler RA, Gill JC, Brabant CP, Mitchell ME, Nugent M, Simpson P, Tweddell JS, Ghanayem NS. Thromboelastography in the assessment of bleeding following surgery for congenital heart disease. World J Pediatr Congenit Heart Surg. 2012 Oct 1;3(4):433-8. doi: 10.1177/2150135112447540. PMID 23804904
- [Result] Williams GD, Bratton SL, Riley EC, Ramamoorthy C. Coagulation tests during cardiopulmonary bypass correlate with blood loss in children undergoing cardiac surgery. J Cardiothorac Vasc Anesth. 1999 Aug;13(4):398-404. doi: 10.1016/s1053-0770(99)90210-0. PMID 10468251
- [Result] Chew MS, Brandslund I, Brix-Christensen V, Ravn HB, Hjortdal VE, Pedersen J, Hjortdal K, Hansen OK, Tonnesen E. Tissue injury and the inflammatory response to pediatric cardiac surgery with cardiopulmonary bypass: a descriptive study. Anesthesiology. 2001 May;94(5):745-53; discussion 5A. doi: 10.1097/00000542-200105000-00010. PMID 11388523
- [Result] Paparella D, Yau TM, Young E. Cardiopulmonary bypass induced inflammation: pathophysiology and treatment. An update. Eur J Cardiothorac Surg. 2002 Feb;21(2):232-44. doi: 10.1016/s1010-7940(01)01099-5. PMID 11825729
- [Result] Bando K, Vijay P, Turrentine MW, Sharp TG, Means LJ, Ensing GJ, Lalone BJ, Sekine Y, Szekely L, Brown JW. Dilutional and modified ultrafiltration reduces pulmonary hypertension after operations for congenital heart disease: a prospective randomized study. J Thorac Cardiovasc Surg. 1998 Mar;115(3):517-25; discussion 525-7. doi: 10.1016/S0022-5223(98)70313-7. PMID 9535437
- [Result] Huang H, Yao T, Wang W, Zhu D, Zhang W, Chen H, Fu W. Continuous ultrafiltration attenuates the pulmonary injury that follows open heart surgery with cardiopulmonary bypass. Ann Thorac Surg. 2003 Jul;76(1):136-40. doi: 10.1016/s0003-4975(03)00264-9. PMID 12842527
- [Result] Forman KR, Wong E, Gallagher M, McCarter R, Luban NL, Massaro AN. Effect of temperature on thromboelastography and implications for clinical use in newborns undergoing therapeutic hypothermia. Pediatr Res. 2014 May;75(5):663-9. doi: 10.1038/pr.2014.19. Epub 2014 Feb 12. PMID 24522100